CLINICAL TRIAL: NCT05097300
Title: Tratamiento de la Cefalea Tensional Mediante técnicas de Tejido Blando VS técnicas de estimulación Del Vago.
Brief Title: Treatment of Tension Headache Using Soft Tissue Techniques VS Vagus Stimulation Techniques.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lucia Trullenque Espallargas (Other)
Responsible Party: Sponsor-Investigator, Lucia Trullenque Espallargas, STUDIENT, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIM/2021/1/017
Record Dates: First submitted 2021-09-14; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Chronic Tension-Type Headache; Episodic Tension-Type Headache
Keywords: Tension type headache; Manual therapy; Vagus nerve stimulation
MeSH Terms: conditions — Tension-Type Headache | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy and vagus nerve stimulation group (Experimental): Patients will recibe 4 sessions, each of the duration of 20 minutes. Manual therapy consist in: suboccipital inhibition (during 10 minutes) and ischemic pressure and passive stretching of three muscles (superior trapezius, temporal muscle and sternocleidomastoid muscle). Vagus nerve stimulation will be performed through a diaphragmatic breathing exercise, during 5 minutes, adding neural tension of median nerve.
  Interventions: Other: Suboccipital inhibition; Other: Ischemic pressure; Other: Passive stretching; Other: Diaphragmatic breathing exercice
- Manual therapy group (Active Comparator): Patients will recibe 4 sessions, each of the duration of 20 minutes. Manual therapy consist in: suboccipital inhibition (during 10 minutes) and ischemic pressure and passive stretching of three muscles (superior trapezius, temporal muscle and sternocleidomastoid muscle).
  Interventions: Other: Suboccipital inhibition; Other: Ischemic pressure; Other: Passive stretching

INTERVENTIONS:
Other: Suboccipital inhibition — The therapist will place his hands under the patient's head, making contact with the suboccipital muscles in the region of the posterior arch of the atlas, applying progressive and deep pressure. This pressure will be maintained for 10 minutes
Other: Ischemic pressure — Pressures will be made on the temporal, superior trapezius, masseter and sternocleidomastoid muscles. Physical therapist will apply gradual sustained finger pressure to the muscle's active trigger points for 5-15 seconds. The therapist will begin with light firm pressure and gradually increase the pressure until the patient feels a "moderate but bearable" level of pain (corresponding to a level 7 on a pain scale of 1 to 10 levels where 1 indicates no pain and 10 is excruciating pain). Pressure will remain at this level until pain levels decrease to level 3. The therapist will repeat this procedure approximately 3-4 times over a 90 second period.
Other: Passive stretching — Passive stretches will be applied to each muscle 2 times for 30 seconds, they will be performed slowly at the rate of the patient's normal breathing and checking that no compensations appear.
Other: Diaphragmatic breathing exercice — To perform diaphragmatic breaths, there will first be an education on how to do them. The patient will lie supine, with the hips and knees semi-flexed. The therapist will ask you to place one hand on your chest and one on your abdomen. Successively, it will ask you to take a few deep breaths, inhaling through your nose for 2 seconds and exhaling through your mouth, with your lips pursed (almost closed) for 4 seconds, helping you to maintain the rhythm of your breath by counting out loud. The patient should note that during inspiration his hand on top of the chest does not rise (the chest remains still) and during expiration that his hand on top of the abdomen goes down (the abdomen sinks).
  Arms: Manual therapy and vagus nerve stimulation group

SUMMARY:
A treatment based on manual therapy and vagus nerve stimulation is more effective than manual therapy only to reduce frequency, intensity and pressure pain threshold in patients with tension type headache.

DETAILED DESCRIPTION:
Participants will be randomly assigned to two groups:

* Experimental group, to which soft tissue techniques and vagus nerve stimulation techniques will be applied.
* Control group, to which only soft tissue techniques are applied. Treatment will consist of four sessions, with an interval of seven days between them, for both study groups. Each session with a duration of 20 minutes for both groups.

In the control group, treatment using soft techniques will consist of the application of manual techniques that have already been shown to have some efficacy in other studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with episodic or chronic tension type headache

Exclusion Criteria:

* Pregnant women
* Patients who have received in the previous 3 months some type of treatment for headache
* Recent history of syncope or seizures
* Heart / cardiovascular disease
* Electrical or neurostimulation devices
* History of intracranial / carotid aneurysm or bleeding; brain tumors / lesions; significant head trauma.
* Change in prophylactic medication type or dose <1 month before the intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity | Day 1 (before the intervention), Day 28 (after the last intervention), Day 56 (4 weeks after the last intervention).
  The strength with which the participants subjectively feel their headache. It will be measured with the following degrees: mild, moderate or severe.
  The Headache Disability Inventory will be used to measure pain intensity.

SECONDARY OUTCOMES:
Change in Headache frequency | Day 1 (before the intervention), Day 28 (after the last intervention), Day 56 (4 weeks after the last intervention).
  The number of headache episodes experienced by the participant in the 30-day time interval (once a month, more than once and less than 4 times a month, and once a week).
  The Headache Disability Inventory will be used to measure headache frequency.
Change in Impact of pain | Day 1 (before the intervention), Day 28 (after the last intervention), Day 56 (4 weeks after the last intervention).
  The impact of pain refers to how much pain affects the patient in the activities of his daily life.
  It will be measured through 25 items of the Headache Disability Inventory.
Change in Pain threshold | Day 1 (before the intervention), Day 28 (after the last intervention).
  Amount of pressure needed to change the patient's sensation from pressure to pain. It will be measured with an algometer, in Newton.
Change in Cervical Range of Motion | Day 1 (before the intervention), Day 28 (after the last intervention).
  It will be measured in degrees, through a cervical goniometer. The patient will be placed in a sitting position. The movements to be measured will be: flexion, whose expected amplitude is 80º; extension with an expected amplitude of 80º; rotations with an expected amplitude of 80º and inclinations with an expected amplitude of 40º.

CONTACTS AND LOCATIONS:
Overall Officials: ALEJANDRO FERRAGUT, DOCTOR, Principal Investigator — Universidad Alcalá de Henares
Locations (2):
- Spain (2):
  - Fisioterapia FIMA clinic, Madrid
  - Facultad de Enfermería y fisioterapia, Universidad Alcalá de Henares, Madrid

IPD SHARING:
Plan to Share IPD: No